CLINICAL TRIAL: NCT00350090
Title: A Pilot Study to Evaluate the Response Rate of PROCRIT (Epoetin Alfa) at 40,000 Units Once Weekly in Anemic Cancer Patients Not Receiving Chemotherapy
Brief Title: A Study to Assess the Response Rate of PROCRIT (Epoetin Alfa) Given at a Dose of 40,000 Units Once a Week to Cancer Patients With Anemia Who Are Not Receiving Chemotherapy.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped early due to slow enrollment.
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005113
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; Neoplasms; Hemoglobin values
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of PROCRIT (Epoetin alfa) administered at 40,000 Units weekly in cancer patients that are not receiving chemotherapy or radiation therapy.

DETAILED DESCRIPTION:
This is an open-label (both the researcher and the patient in the study know the treatment that is being given), non-randomized, multi-center pilot study with the objective to investigate the efficacy of PROCRIT (Epoetin alfa) with regard to hematopoietic response when administered at 40,000 Units subcutaneously (under the skin) once per week in anemic patients with cancer not receiving chemotherapy or radiation therapy. Hematological laboratory tests (hemoglobin and hematocrit), vital signs (blood pressure) and occurrence and severity of adverse events will be assessed throughout the study. Patients will receive a PROCRIT (Epoetin alfa) injection (40,000 Units per injection) under the skin once every week for a maximum of 13 weeks. Doses may be reduced depending on the patients' hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin value of less than or equal to 11 g/dL unrelated to transfusion
* Patients must not be receiving or planning to receive chemotherapy or radiotherapy within the 16-week study period. However, patients receiving hormonal therapy or non-myelosuppressive therapies are allowable
* Female patients with reproductive potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* Uncontrolled hypertension
* History (within 6 months) of uncontrolled cardiac arrhythmias, or history of pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic coagulation disorder
* Transfusion within 28 days prior to first dose
* Planned chemotherapy or radiation during study and no prior chemotherapy within 8 weeks or radiation within 4 weeks of study entry
* No prior treatment with Epoetin alfa or any other erythropoietic agent within the previous two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2002-09; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Hematologic response in terms of hemoglobin and transfusion requirements where hemoglobin response is characterized as minor > 1g/dL Hb increase or major > 2g/dL Hb increase.

SECONDARY OUTCOMES:
Secondary efficacy variables will include the effects of PROCRIT (Epoetin alfa) on transfusion requirements and on Quality of Life as measured by the Linear Analog Scale Assessment (LASA) tool.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Shasha D, Williams D. Weekly epoetin alfa treatment of anemia in patients with cancer not undergoing therapy. J Support Oncol. 2006 Mar;4(3):129-35. PMID 16553139
- See also: A Pilot Study to Evaluate the Response Rate of PROCRIT (Epoetin alfa) at 40,000 Units Once Weekly in Anemic Cancer Patients Not Receiving Chemotherapy or Radiation Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=928&filename=CR005113_CSR.pdf